CLINICAL TRIAL: NCT04944576
Title: Observational Multicenter Prospective Clinical Study on the Total Ankle Prosthesis, EasyMove®, Evaluating Safety and Performance up to 5 Years of Follow-up
Brief Title: Observational Study to Evaluate Safety and Performance of the Total Ankle Prosthesis, EasyMove®
Status: Active, not recruiting | Type: Observational
Sponsor: FH ORTHO (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-42; 2020-A03401-38 (Registry Identifier: French registry related to the ANSM (ID-RCB))
Record Dates: First submitted 2021-06-14; First posted 2021-06-29 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Ankle Injuries and Disorders
MeSH Terms: conditions — Ankle Injuries; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Total Ankle Prosthesis, EasyMove® — Patients who will be implanted with a total ankle prosthesis, EasyMove.

SUMMARY:
This study is a post-market clinical follow-up conducted in order to collect long-term data on safety and performance of the EasyMove prosthesis, which is intended to be implanted in case of total ankle replacement, when used in real life conditions according to the instructions for use.

DETAILED DESCRIPTION:
The primary objective is to evaluate the safety of the total ankle prosthesis, EasyMove, up to five years of follow-up.

The secondary objectives are to evaluate both the safety and the performance of the total ankle prosthesis, EasyMove, up to five years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient implanted with the studied device according to the instructions for use, for primary surgery in patients with ankle joints damaged by severe rheumatoid, post-traumatic or degenerative arthritis
* Adult patient (≥18 years old)
* Patient who received an information form and is willing to participate in the study

Exclusion Criteria:

* Contraindications listed in the instructions for use
* Patient who is not able to express his/her non opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from participating centres will be enrolled as part of their clinical routine care.
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2029-09-13 (Estimated); Study Completion 2029-09-13 (Estimated)

PRIMARY OUTCOMES:
Revision rate | Up to 5 years of follow-up
  Revision rate of the implant for aseptic loosening.

SECONDARY OUTCOMES:
Functional outcomes evaluation such as pain and mobility | preop, 4-6 weeks postop, 1 year postop, 2 years postop, 5 years postop
  Functional ouctomes will be evaluated through the AOFAS score. This score is comprised of nine questions covering three categories: pain (40 points), function (50 points) and alignment (10 points). These are all scored together for a total of 100 points. The higher the score, the better the patient outcome. AOFAS is a clinician reporting tool that required both patient and provider participation to be fully complete. The AOFAS score will be compared to its MCID at each follow-up visit. The MCID will be calculated based on the distribution-based MCID method.
Functional outcomes evaluation such as mobility | preop, 1 year postop, 2 years postop, 5 years postop
  Functional ouctomes will be evaluated through the FAAM score. This score is a 29-item questionnaire divided into two subscales: 21-item Activities of Daily Living Subscale and 8-item Sports Subscale. Item score totals, which range from 0 to 84 for the Activities of Daily Living subscale and 0 to 32 for the Sports subscale, are transformed to percentage scores. The higher the score, the better the patient outcomes. It is a self-report outcome instrument. The FAAM score will be compared to its MCID at each follow-up visit. The Minimal Clinically Important Difference (MCID) of the Foot and Ankle Ability Measure (FAAM) at 1 year of follow-up compared to the theorical MCID retrieved in the literature (MCID = 31.2 (sd=25.3, superiority comparison)). For the following follow-up, the MCID will be calculated based on the distribution-based MCID method.
Functional outcomes evaluation such as mobility | preop, 4-6 weeks postop, 1 year postop, 2 years postop, 5 years postop
  Functional ouctomes will be evaluated through clinical data such as the range of motion.
Health status outcomes evaluation such as pain | preop, 4-6 weeks postop, 1 year postop, 2 years postop, 5 years postop
  Health status outcomes will be evaluated through a visual analogue scale to measure pain.
Health status outcomes evaluation such as quality of life | preop, 1 year postop, 2 years postop, 5 years postop
  Health status outcomes will be evaluated through the SF-12 questionnaire to measure the quality of life. It is a self-reported outcome measure, composed of 12 questions. It provides an eight-scale profile of functional health and wellbeing, as well as two psychometrically based physical and mental health summary measures, scored on a T-score metric. The higher the score, the better the patient outcomes. The SF-12 score will be compared to its MCID at each follow-up visit. The MCID will be calculated based on the distribution-based MCID method.
Radiological data evaluation | preop, 4-6 weeks postop, 1 year postop, 2 years postop, 5 years postop
  Radiological data results such as the postion of the implant, lucency, calcification will be evaluated.
Rate of complications | perop, 4-6 weeks postop, 1 year postop, 2 years postop, 5 years postop
  All complications will be gathered from the intervention up to 5 years of follow-up.

CONTACTS AND LOCATIONS:
Locations (6):
- France (5):
  - Chu Brest, Brest
  - CH Raymond-Poincaré, Garches
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Clinique Victor HUGO, Paris
  - Clinique Jouvenet, Paris
- Centre hospitalier universitaire vaudois, Lausanne, Switzerland